CLINICAL TRIAL: NCT02163070
Title: Effect of Vitamin E Fortified Whey Drink on Nutritional Status, Inflammatory Markers and Oxidative Stress in Hemodialysis Patients
Brief Title: Effect of Vitamin E Fortified Whey Drink on Nutritional, Inflammatory and Oxidative Markers in Hemodialysis Patients
Acronym: EVEWD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mohammad Hassan Eftekhari (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Mohammad Hassan Eftekhari, professor. PhD, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91-6424
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Kidney Disease
Keywords: whey protein; malnutrition; oxidative stress; hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Malnutrition | interventions — Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- whey drink (Experimental): consumption of 220 milliliters of whey drink three times a week,
  Interventions: Dietary Supplement: whey drink,
- whey drink fortified with vitaminE (Experimental): consumption of 220 milliliters of whey drink fortified with 400 milligrams of vitamin E three times a week,
  Interventions: Dietary Supplement: whey drink fortified with vitaminE
- vitaminE (Experimental): consumption of 400 milligrams of vitamin E three times a week,
  Interventions: Dietary Supplement: vitamin E
- D- control (No Intervention): control group: no intervention,

INTERVENTIONS:
Dietary Supplement: whey drink, — consumption of 220 milliliters of whey drink three times a week,
  Arms: whey drink
Dietary Supplement: whey drink fortified with vitaminE — consumption of 220 milliliters of whey drink fortified with 400 milligrams of vitamin E three times a week,
  Arms: whey drink fortified with vitaminE
Dietary Supplement: vitamin E — consumption of 400 milligrams of vitamin E three times a week,
  Arms: vitaminE

SUMMARY:
The purpose of the study is to evaluate the effect of vitamin E fortified whey drink on nutritional status, inflammatory markers and oxidative stress in hemodialysis patients

DETAILED DESCRIPTION:
The aim of this interventional study was to evaluate the effect of vitamin E fortified whey drink on nutritional status, inflammatory markers and oxidative stress in hemodialysis patients. 92 hemodialysis patients were selected for the study. Inclusion criteria included: mean age of 17-65 years old; having mild, moderate or severe malnutrition based on the SGA (subjective global assessment) assessment; being dialyzed at least 2 times a week for 3 months. Exclusion criteria included: hospitalization in the last month; active infection; using immunosuppressant drugs or multi-vitamins; pregnancy. The Ethics Committee of Shiraz University of Medical Sciences reviewed and approved the protocol of this study.Informed consent were signed by all of them for participating in the study. Weight and height of the patients were recorded for BMI (body mass index) calculation. Then, all of the patients were assigned into 4 groups:

1. consumption of 220 milliliters of whey drink three times a week,
2. consumption of 220 milliliters of whey drink fortified with 400 milligrams of vitamin E three times a week,
3. consumption of 400 milligrams of vitamin E three times a week,
4. control group: no intervention. Patients were followed for 2 months. At the beginning and the end of the 2-month intervention period, 10 milliliters of blood were taken from all of the patients and nutritional status of the patients were assessed as the primary outcome. Serum levels of malondialdehyde, c-reactive protein, albumin, transferrin and lipoproteins were also measured. SGA, MIS and SF-12 questionnaires were filled for all of the patients at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* mean age of 17-65 years old;
* having mild, moderate or severe malnutrition based on the SGA (subjective global assessment) assessment;
* be dialyzed at least 2 times a week for 3 months

Exclusion Criteria:

* hospitalization in the last month;
* active infection;
* using immunosuppressant drugs or multi-vitamins;
* pregnancy, consuming whey or soy products

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
malnutrition (based on SGA assessment) | 2 months (8 weeks)
Malnutrition inflammation score | 2 months (8 weeks)

SECONDARY OUTCOMES:
serum interleukin-6 | 2 months (8 weeks)
serum C-reactive protein | 2 months (8 weeks)
serum albumin | 2 months (8 weeks)
serum HDL-c | 2 months (8 weeks)
serum total cholesterol | 2 months (8 weeks)
serum triglyceride | 2 months (8 weeks)
serum transferrin | 2 months (8 weeks)
serum malondialdehyde | 2 months (8 weeks)
BUN (blood urea nitrogen) | 2 months (8 weeks)
serum creatinine | 2 months (8 weeks)
serum calcium | 2 months (8 weeks)
serum phosphate | 2 months (8 weeks)
quality of life | 2 months (8 weeks)
weight | 2 months (8 weeks)
height | 2 months (8 week)
Body mass index | 2 months (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hassan Eftekhari, professor, Study Director — Shiraz University of Medical Sciences

REFERENCES:
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133